CLINICAL TRIAL: NCT02100670
Title: A Clinical Study to Assess the Efficacy and Onset of Pain Relief of Topical MFC51123 Diclofenac-Menthol Gel Versus Controls in Ankle Sprain
Brief Title: A Multicenter Efficacy Study of a Diclofenac+Menthol Gel in Subjects With Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202179; RH01805 (Other: GSK)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac; Menthol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1% diclofenac sodium plus 3% menthol (Experimental): 1% diclofenac sodium plus 3% menthol gel supplied in 30 gram (g) tubes sufficient for each subject to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
  Interventions: Drug: 1% diclofenac sodium plus 3% menthol
- 1% diclofenac sodium plus 0.09% menthol (Experimental): 1% diclofenac sodium plus 0.09% menthol gel supplied in 30g tubes sufficient for each subject to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
  Interventions: Drug: 1% diclofenac sodium plus 0.09% menthol
- 3% menthol (Experimental): 3% menthol gel supplied in 30g tubes sufficient for each subject to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
  Interventions: Drug: 3% menthol
- Placebo with 0.09% menthol gel (Placebo Comparator): Placebo with 0.09% menthol gel supplied in 30g tubes sufficient for each subject to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
  Interventions: Drug: Placebo with 0.09% menthol gel

INTERVENTIONS:
Drug: 1% diclofenac sodium plus 3% menthol — To be applied four times daily for 10 days.
  Arms: 1% diclofenac sodium plus 3% menthol
Drug: 1% diclofenac sodium plus 0.09% menthol — To be applied four times daily for 10 days.
  Arms: 1% diclofenac sodium plus 0.09% menthol
Drug: 3% menthol — To be applied four times daily for 10 days.
  Arms: 3% menthol
Drug: Placebo with 0.09% menthol gel — To be applied four times daily for 10 days.
  Arms: Placebo with 0.09% menthol gel

SUMMARY:
This Phase III pivotal efficacy study will assess efficacy and onset of pain relief of MFC51123 gel vs. placebo and MFC51123 gel vs. 1% diclofenac gel and 3% menthol gel in participants with an ankle sprain to support topical MFC51123 gel registration.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, repeat-dose, placebo-controlled, parallel-group trial in participants with ankle sprain. Eligible participants will be randomly assigned to one of four treatment groups (1% diclofenac plus 3% menthol gel, 1% diclofenac plus 0.09% menthol gel, 3% menthol gel or placebo gel with 0.09% menthol). Treatment will be self-administered by participants four times daily on an out-patient basis. Participants will rate pain intensity score (NRS) at rest and on movement, pain relief score (PRS) and cooling and soothing sensations. After leaving the clinic, participants will continue to complete scheduled pain intensity and pain relief assessments and answer questions about cooling sensation by answering questions in a paper diary card. The investigator (or designee) will measure the ankle swelling via the 'figure-of-eight' method on treatment Days 1 (at Baseline), 3, 7 and 10.

Participants will continue treatment until they are pain free or for up to 10 days, whichever occurs first. At the end of the treatment, participants will be assessed for function of the injured joint by the investigator. In addition, the participants will evaluate treatment satisfaction, sensory features of the gel and provide a global assessment of the treatment by using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-65 years
* Good general and mental health
* Grade I or Grade II acute sprain of the lateral ankle within 24 hours of Visit 1, a pain intensity score of the ankle sprain that is ≥ 5 as measured on an 11-point numerical rating scale, and a peri-malleolar edema (sub-malleolar perimeter difference of ≥ 20mm between injured and uninjured ankle
* Females of child-bearing age practicing a reliable method of contraception

Exclusion Criteria:

* Pregnant or breast-feeding females
* If participant has treated the ankle sprain with treatment such as oral or other topical pain relief medications, massage or physical therapy since experiencing the ankle sprain
* Acute or chronic pain disorders, which may confound the study pain evaluations
* Participant has has injury to both ankles or to both medial and lateral ligaments of the same ankle
* Known or suspected hypersensitivity, allergy, intolerance or contraindication to the use of any of the study medications
* Participant has a medical history of renal or hepatic disease, a current active peptic ulcer or a history of upper gastrointestinal bleeding or perforation related to previous NSAID therapy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2013-11-01; Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - PAREXEL International - Sites in Germany, Berlin
  - PAREXEL International, LLC, Berlin
  - pro scientia med im MARE Klinikum, Kiel

REFERENCES:
- [Derived] Lai PM, Collaku A, Reed K. Efficacy and safety of topical diclofenac/menthol gel for ankle sprain: A randomized, double-blind, placebo- and active-controlled trial. J Int Med Res. 2017 Apr;45(2):647-661. doi: 10.1177/0300060517700322. Epub 2017 Mar 27. PMID 28345425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 16 centers in Germany.
Pre-assignment Details: A total of 388 participants were screened, out of which 385 were randomized, 3 did not meet the study criteria. Of the 385 participants randomized, 360 participants completed the study, 25 did not complete the study.
Groups:
- 1% Diclofenac Sodium+3% Menthol: 1% diclofenac sodium with 3% menthol gel was supplied in 30 gram (g) tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- 1% Diclofenac Sodium: 1% diclofenac sodium with 0.09% methanol gel was supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- 3% Menthol: 3% menthol gel was supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- Placebo: Placebo with 0.09% methanol gel was supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
Period: Overall Study
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Started | 118 | 113 | 78 | 76
Completed | 105 | 106 | 74 | 75
Not Completed | 13 | 7 | 4 | 1
Not completed — Adverse Event | 10 | 3 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 1 | 1 | 0
Not completed — No swelling no pain | 1 | 0 | 0 | 0
Not completed — Poor Efficacy | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 381 participants were included in safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo | Total
Number analyzed (Participants) | 117 | 112 | 77 | 75 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.4 (11.83) | 32.1 (11.40) | 33.8 (12.15) | 33.2 (11.63) | 32.8 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 39 | 35 | 165
  Male | 67 | 71 | 38 | 40 | 216

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Day 1 to Day 3 (AUC1-3 Days) of Pain Intensity(PI) on Movement for Diclofenac/Methanol Gel and Placebo Gel
Description: AUC of PI on movement was measured by a numerical rating scale (NRS) during the 48 hour time interval from Day 1 to 3. AUC1-3 day was calculated based on trapezoidal method. Pain intensity was measured in NRS scale from 0 (no pain) to 10 (extreme pain). Participants assessed the severity of ankle pain using the NRS scale at baseline (prior to treatment) and at 10, 30 minutes and 1, 4, 6, 12, 18 and 24 hours after the first dose of treatment and twice daily after dosing.
Time Frame: up to 72 hours
Population: Intent-to-Treat (ITT) population included all participants who fulfilled all the study entry criteria, received the study treatment and had at least one post-baseline efficacy assessment. This analysis was conducted on ITT population.
Measure: Mean (Standard Deviation); unit: NRS Score (0 - 10 scale) * hrs
Groups:
- 1% Diclofenac Sodium Plus (+) 3% Menthol: 1% diclofenac sodium+3% menthol gel was supplied in 30 gram (g) tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- Placebo: Placebo gel was supplied in 30g tubes for each participant to apply 4g of gel topically to the injured ankle region four times daily for up to 10 days.
Arm/Group | 1% Diclofenac Sodium Plus (+) 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 75
NRS Score (0 - 10 scale) * hrs | 276.97 (111.356) | 282.88 (100.958)
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium Plus (+) 3% Menthol vs Placebo; Test type: Superiority or Other; p = 0.4144, ANCOVA — P-value from multiple comparisons using t-test in Proc Mixed; Least squares (LS) means from mixed model analysis of covariance with treatment, site as fixed effects, pain intensity at baseline as a covariates; Difference of LS mean = -9.23, 95% CI 2-sided [-31.45 to 12.98] — Difference of LS mean of first named treatment minus second named treatment. Lower values of LS mean favours a better response because of lower pain intensity over time. 95% Confidence intervals of difference between LS means

2. Secondary Outcome: AUC1-3 Days of PI on Movement for Diclofenac Sodium + Methanol, Diclofenac, Methanol and Placebo
Description: as for outcome 1
Time Frame: up to 72 hours
Population: ITT population included all participants who fulfilled all the study entry criteria, received the study treatment and had at least one post-baseline efficacy assessment. This analysis was conducted on ITT population.
Measure: Mean (Standard Deviation); unit: NRS Score (0 - 10 scale) * hrs
Groups:
- 1% Diclofenac Sodium+3% Menthol: 1% diclofenac sodium+3% menthol gel was supplied in 30 gram (g) tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
NRS Score (0 - 10 scale) * hrs | 276.97 (111.356) | 261.11 (96.791) | 272.65 (118.196) | 282.88 (100.958)
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium+3% Menthol vs 1% Diclofenac Sodium; Test type: Superiority or Other; p = 0.8761, ANCOVA — P-value from multiple comparisons using t-test in Proc Mixed; [statistical method as in outcome 1, analysis 1]; LS mean difference = 1.58, 95% CI 2-sided [-18.34 to 21.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1% Diclofenac Sodium+3% Menthol vs 3% Menthol; Test type: Superiority or Other; p = 0.8164, ANCOVA — P-value from multiple comparisons using t-test in Proc Mixed; [statistical method as in outcome 1, analysis 1]; LS mean difference = 2.61, 95% CI 2-sided [-19.46 to 24.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 1% Diclofenac Sodium vs 3% Menthol; Test type: Superiority or Other; p = 0.9279, ANCOVA — P-value from multiple comparisons using t-test in Proc Mixed; [statistical method as in outcome 1, analysis 1]; LS mean difference = 1.03, 95% CI 2-sided [-21.27 to 23.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 1% Diclofenac Sodium vs Placebo; Test type: Superiority or Other; p = 0.3442, ANCOVA — P-value from multiple comparisons using t-test in Proc Mixed; [statistical method as in outcome 1, analysis 1]; LS mean difference = -10.81, 95% CI 2-sided [-33.26 to 11.64] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Pain Intensity Difference (PID) on Movement
Description: PID on movement, calculated as PI at a given time 't' (after walking 5 steps on a flat surface) subtracted by the PI at baseline.
  Participants assessed the severity of ankle pain (PI) using the NRS scale from 0 (no pain) to 10 (extreme pain). PI was measured at baseline (prior to treatment) and at 10, 30 minutes (min.) and 1, 4, 6, 12, 18 and 24 hours after the first dose of treatment and twice daily after dosing.
Time Frame: Baseline to 10 days
Population: ITT population included all participants who fulfilled all the study entry criteria, received the study treatment and had at least one post-baseline efficacy assessment. This analysis was conducted on ITT population. n is number of participants analyzed for respective time point for this outcome.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
score on scale
  PI at Baseline (n=117, 112, 77, 75) | 7.8 (1.55) | 7.4 (1.44) | 7.8 (1.60) | 7.7 (1.47)
  PID at 10 min. (n=117, 112, 77, 75) | 0.23 (1.078) | 0.19 (0.855) | 0.29 (0.886) | 0.32 (1.129)
  PID at 30 min. (n=117, 112, 77, 75) | 0.44 (1.302) | 0.36 (0.967) | 0.49 (0.868) | 0.55 (1.464)
  PID at 1 hour (n=117, 112, 77, 75) | 0.56 (1.348) | 0.50 (1.022) | 0.64 (1.146) | 0.64 (1.521)
  PID at 4 hour (n=117, 112, 77, 75) | 0.71 (1.640) | 0.48 (1.057) | 0.79 (1.128) | 0.69 (1.414)
  PID at 6 hour (n=117, 112, 77, 75) | 0.79 (1.706) | 0.67 (1.094) | 0.91 (1.227) | 0.87 (1.554)
  PID at 12 hour (n= 117, 112, 77, 75) | 0.84 (1.692) | 0.99 (1.411) | 1.17 (1.542) | 0.95 (1.550)
  PID at 18 hour (n=117, 112, 77, 75) | 1.19 (1.707) | 1.32 (1.409) | 1.44 (1.751) | 1.16 (1.661)
  PID at 24 hour (n=117, 112, 77, 75) | 1.62 (1.866) | 1.58 (1.505) | 1.75 (1.808) | 1.53 (1.639)
  PID at 36 hour (n=117, 112, 77, 75) | 1.59 (1.899) | 1.65 (1.592) | 1.55 (1.818) | 1.32 (1.702)
  PID at 48 hour (n=117, 112, 77, 75) | 1.91 (1.914) | 2.01 (1.562) | 2.04 (1.874) | 1.92 (1.937)
  PID at 60 hour (n=117, 112, 77, 75) | 2.41 (1.917) | 2.26 (1.659) | 2.56 (1.963) | 2.05 (1.888)
  PID at 72 hour (n=117, 112, 77, 75) | 2.55 (1.989) | 2.42 (1.631) | 2.55 (1.977) | 2.28 (1.935)
  PID at 84 hour (n=113, 107, 75, 75) | 2.84 (1.883) | 2.68 (1.686) | 3.08 (1.916) | 2.68 (2.008)
  PID at 96 hour (n=112, 107, 75, 74) | 3.10 (1.865) | 2.78 (1.890) | 3.03 (2.027) | 2.78 (1.882)
  PID at 108 hour (n=112, 107, 75, 74) | 3.34 (1.980) | 3.01 (1.751) | 3.48 (1.989) | 3.18 (1.996)
  PID at 120 hour (n=111, 107, 74, 74) | 3.38 (1.864) | 3.17 (1.871) | 3.35 (2.044) | 3.14 (1.947)
  PID at 132 hour (n=110, 107, 74, 74) | 3.70 (1.961) | 3.53 (1.824) | 3.72 (1.913) | 3.47 (2.042)
  PID at 144 hour (n=110, 107, 74, 74) | 3.76 (2.058) | 3.78 (1.870) | 3.68 (1.994) | 3.59 (1.979)
  PID at 156 hour (n=109, 107, 74, 74) | 4.17 (2.115) | 4.05 (1.870) | 3.95 (1.999) | 3.88 (2.158)
  PID at 168 hour (n=105, 104, 73, 74) | 4.26 (2.103) | 4.11 (1.935) | 3.90 (2.122) | 3.95 (2.067)
  PID at 180 hour (n=105, 104, 73, 72) | 4.58 (2.065) | 4.45 (1.980) | 4.37 (1.933) | 4.08 (2.121)
  PID at 192 hour (n=101, 102, 71, 72) | 4.55 (2.081) | 4.59 (1.916) | 4.21 (2.197) | 4.22 (2.023)
  PID at 204 hour (n=101, 100, 71, 72) | 5.17 (2.020) | 4.94 (1.984) | 4.87 (1.999) | 4.56 (2.122)
  PID at 216 hour (n=95, 100, 69, 72) | 5.28 (2.239) | 5.21 (2.100) | 4.87 (2.029) | 4.78 (1.987)
  PID at 228 hour (n=95, 100, 69, 72) | 5.71 (2.292) | 5.62 (2.068) | 5.28 (2.071) | 5.01 (2.113)
  PID at 240 hour (n=32, 43, 22, 42) | 5.56 (2.961) | 5.44 (2.196) | 5.41 (2.282) | 5.60 (1.951)

4. Secondary Outcome: PID at Rest
Description: PID at rest was calculated as PI at a given time point't' (at rest) subtracted by the PI at baseline. Participants assessed the severity of ankle pain (PI) using the NRS scale from 0 (no pain) to 10 (extreme pain).
  PI was measured at baseline (prior to treatment) and at 10, 30 minutes and 1, 4, 6, 12, 18 and 24 hours after the first dose of treatment and twice daily after dosing.
Time Frame: Baseline to 10 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 3% Menthol: 3% menthol gel supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
score on a scale
  PI at Baseline (n=117, 112, 77, 75) | 7.8 (1.55) | 7.4 (1.44) | 7.8 (1.60) | 7.7 (1.47)
  PID at 10 min. (n=117, 112, 77, 75) | 0.34 (1.146) | 0.43 (1.145) | 0.17 (0.715) | 0.25 (1.175)
  PID at 30 min. (n=117, 112, 77, 75) | 0.56 (1.185) | 0.45 (1.314) | 0.32 (0.818) | 0.44 (1.328)
  PID at 1 hour (n=117, 112, 77, 75) | 0.64 (1.283) | 0.62 (1.187) | 0.48 (0.940) | 0.41 (1.620)
  PID at 4 hour (n=117, 112, 77, 75) | 0.62 (1.413) | 0.53 (1.115) | 0.66 (1.071) | 0.43 (1.678)
  PID at 6 hour (n= 117, 112, 77, 75) | 0.68 (1.473) | 0.62 (1.180) | 0.75 (1.183) | 0.53 (1.554)
  PID at 12 hour (n= 117, 112, 77, 75) | 0.76 (1.501) | 0.86 (1.432) | 0.90 (1.429) | 0.68 (1.535)
  PID at 18 hour (n= 117, 112, 77, 75) | 1.03 (1.597) | 1.14 (1.482) | 1.10 (1.594) | 0.85 (1.666)
  PID at 24 hour (n= 117, 112, 77, 75) | 1.32 (1.579) | 1.39 (1.448) | 1.47 (1.535) | 1.13 (1.711)
  PID at 36 hour (n= 117, 112, 77, 75) | 1.20 (1.549) | 1.32 (1.490) | 1.22 (1.635) | 1.09 (1.787)
  PID at 48 hour (n=117, 112, 77, 75) | 1.43 (1.604) | 1.53 (1.464) | 1.51 (1.698) | 1.45 (1.840)
  PID at 60 hour (n= 117, 112, 77, 75) | 1.91 (1.603) | 1.83 (1.593) | 1.88 (1.747) | 1.64 (1.893)
  PID at 72 hour (n= 117, 112, 77, 75) | 1.91 (1.776) | 1.91 (1.545) | 1.86 (1.782) | 1.76 (1.972)
  PID at 84 hour (n= 113, 107, 75, 75) | 2.11 (1.754) | 2.19 (1.655) | 2.19 (1.799) | 2.03 (1.931)
  PID at 96 hour (n= 112, 107, 75, 74) | 2.26 (1.790) | 2.17 (1.707) | 2.23 (1.721) | 2.00 (1.720)
  PID at 108 hour (n=112, 107, 75, 74) | 2.46 (1.795) | 2.43 (1.833) | 2.48 (1.743) | 2.27 (1.889)
  PID at 120 hour (n= 111, 107, 74, 74) | 2.59 (1.836) | 2.48 (1.750) | 2.30 (1.856) | 2.09 (1.917)
  PID at 132 hour (n= 110, 107, 74, 74) | 2.76 (1.877) | 2.78 (1.819) | 2.68 (1.873) | 2.49 (1.967)
  PID at 144 hour (n= 110, 107, 74, 74) | 2.77 (1.989) | 2.77 (1.789) | 2.59 (1.965) | 2.49 (1.918)
  PID at 156 hour (n= 109, 107, 74, 74) | 3.06 (2.011) | 3.11 (1.755) | 2.77 (1.884) | 2.65 (2.129)
  PID at 168 hour (n= 105, 104, 73, 74) | 3.08 (2.037) | 3.15 (1.805) | 2.75 (1.869) | 2.64 (2.004)
  PID at 180 hour (n= 105, 104, 73, 72) | 3.37 (2.100) | 3.38 (1.871) | 2.95 (1.747) | 2.88 (2.103)
  PID at 192 hour (n= 101, 102, 71, 72) | 3.38 (2.240) | 3.30 (2.067) | 2.90 (1.928) | 3.00 (2.035)
  PID at 204 hour (n= 101, 100, 71, 72) | 3.67 (2.250) | 3.61 (2.030) | 3.37 (1.853) | 3.21 (2.021)
  PID at 216 hour (n= 95, 100, 69, 72) | 3.77 (2.372) | 3.87 (2.028) | 3.22 (2.306) | 3.26 (1.936)
  PID at 228 hour (n= 95, 100, 69, 72) | 4.09 (2.348) | 4.02 (2.074) | 3.64 (2.000) | 3.53 (2.083)
  PID at 240 hour (n= 32, 43, 22, 42) | 3.94 (2.862) | 4.23 (2.010) | 3.36 (2.610) | 3.67 (2.149)

5. Secondary Outcome: Pain Relief Score (PRS)
Description: Pain relief was measured at each time point using a 5-point Pain Relief Scale ranging from 0-4 while at rest (Where: 0- No pain relief; 1- A little or perceptible pain relief; 2- Meaningful pain relief; 3- A lot of relief; 4- Complete relief). Participants assessed the degree of ankle pain relief using the PRS scores at 10, 30 minutes and 1, 4, 6, 12, 18 and 24 hours after the first dose of treatment and twice daily after the first day of treatment.
Time Frame: Day 1 to Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
score on a scale
  At 10 min. (n= 117, 111, 77, 74) | 0.33 (0.616) | 0.29 (0.609) | 0.32 (0.498) | 0.36 (0.610)
  At 30 min. (n=117, 111, 77, 75) | 0.44 (0.635) | 0.36 (0.585) | 0.49 (0.599) | 0.44 (0.683)
  At 1 hour (n=116, 112, 77, 75) | 0.48 (0.625) | 0.46 (0.599) | 0.57 (0.677) | 0.40 (0.717)
  At 4 hour (n= 115, 110, 74, 71) | 0.47 (0.626) | 0.45 (0.552) | 0.51 (0.579) | 0.49 (0.673)
  At 6 hour (n= 109, 105, 70, 69) | 0.50 (0.603) | 0.54 (0.605) | 0.63 (0.618) | 0.45 (0.607)
  At 12 hour (n= 77, 89, 53, 58) | 0.60 (0.591) | 0.72 (0.707) | 0.74 (0.684) | 0.62 (0.745)
  At 18 hour (n= 76, 78, 53, 57) | 0.71 (0.689) | 0.73 (0.715) | 0.83 (0.753) | 0.70 (0.680)
  At 24 hour (n= 111, 105, 72, 72) | 0.79 (0.662) | 0.74 (0.680) | 0.90 (0.754) | 0.81 (0.642)
  At 36 hour (n= 116, 112, 77, 74) | 0.84 (0.709) | 0.84 (0.705) | 0.88 (0.760) | 0.78 (0.781)
  At 48 hour (n= 116, 112, 77, 75) | 0.90 (0.806) | 0.84 (0.651) | 0.99 (0.716) | 0.99 (0.846)
  At 60 hour (n=115, 111, 77, 75) | 1.07 (0.780) | 1.00 (0.714) | 1.16 (0.745) | 0.96 (0.779)
  At 72 hour (n= 114, 109, 75, 74) | 0.93 (0.784) | 1.06 (0.743) | 1.16 (0.806) | 0.97 (0.810)
  At 84 hour (n= 113, 106, 75, 75) | 1.07 (0.810) | 1.00 (0.756) | 1.25 (0.737) | 1.11 (0.746)
  At 96 hour (n= 112, 106, 75, 74) | 1.09 (0.823) | 1.03 (0.762) | 1.01 (0.830) | 1.09 (0.743)
  At 108 hour (n= 111, 105, 75, 74) | 1.18 (0.876) | 1.13 (0.809) | 1.28 (0.894) | 1.15 (0.734)
  At 120 hour (n= 111, 107, 74, 72) | 1.11 (0.918) | 1.14 (0.782) | 1.24 (0.904) | 1.10 (0.772)
  At 132 hour (n= 110, 107, 73, 74) | 1.34 (0.931) | 1.24 (0.878) | 1.34 (0.931) | 1.30 (0.887)
  At 144 hour (n= 110, 107, 74, 73) | 1.21 (1.015) | 1.21 (0.919) | 1.30 (0.947) | 1.27 (0.886)
  At 156 hour (n= 109, 106, 74, 74) | 1.41 (1.011) | 1.30 (1.053) | 1.47 (0.968) | 1.32 (0.952)
  At 168 hour (n= 105, 103, 73, 73) | 1.41 (1.026) | 1.31 (0.990) | 1.34 (1.003) | 1.40 (0.924)

6. Secondary Outcome: Sum of Pain Intensity Difference (SPID)
Description: SPID was calculated as the time weighted sum of pain intensity differences (PID) from 0 to 7 Days. PID was calculated as PI at a given time point 't' subtracted by the PI at baseline. PI was measured on NRS scale from 0 (no pain) to 10 (extreme pain). The possible range of SPID for 0-6 hours was from -60 to 60, for 0-12 hours was from -120 to 120, for 0-1 day was from -240 to 240, for 0-3 days was from -720 to 720, for 0-7 days was from -1680 to 1680. A higher value of SPID indicates greater pain relief.
Time Frame: Baseline to Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
score on a scale
  At 0-6 hours | 4.16 (9.299) | 3.19 (5.862) | 4.72 (6.306) | 4.37 (8.287)
  At 0-12 hours | 9.19 (18.788) | 9.13 (13.284) | 11.74 (14.675) | 10.05 (16.706)
  At 0-1 days | 26.01 (38.722) | 26.54 (28.497) | 30.91 (34.158) | 26.21 (34.877)
  At 1 to 3 days | 101.54 (87.184) | 100.07 (71.085) | 104.26 (83.689) | 90.88 (82.626)
  At 0 to 7 days | 451.12 (265.919) | 452.44 (244.488) | 464.96 (281.243) | 438.45 (287.369)

7. Secondary Outcome: Time of Onset of Pain Relief (TOPR)
Description: TOPR was measured by time when participants reported PRS ≥ 1, i.e. a "little" or "perceptible" pain relief'.
Time Frame: Baseline to 10 days (end of study)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
Hours | 1.03 [0.2 to 157.0] | 4.00 [0.2 to 168.0] | 1.00 [0.2 to 94.3] | 4.00 [0.2 to 187.5]
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium+3% Menthol vs Placebo; Test type: Superiority or Other; p = 0.5404, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.10, 95% CI 2-sided [0.81 to 1.48] — Cox proportional hazard ratio of survival time, i.e. time to reach perceptible pain relief. The 95% confidence intervals of cox proportional hazard ratio
Statistical Analysis 2: Comparison: 1% Diclofenac Sodium+3% Menthol vs 3% Menthol; Test type: Superiority or Other; p = 0.4639, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 0.90, 95% CI 2-sided [0.67 to 1.20] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 1% Diclofenac Sodium+3% Menthol vs 1% Diclofenac Sodium; Test type: Superiority or Other; p = 0.5118, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.09, 95% CI 2-sided [0.84 to 1.43] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Time of Onset of Meaningful Pain Relief (TOMR)
Description: TOMR was measured by time when participants reported PRS ≥ 2, i.e. "some" or "meaningful" pain relief
Time Frame: up to 10 days (end of study)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Groups:
- 1% Diclofenac Sodium+3% Menthol: 1% diclofenac sodium+3% menthol gel was supplied in 30 gram (g) tubes sufficient for each participants to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- 1% Diclofenac Sodium: 1% diclofenac sodium with 0.09% methanol gel was supplied in 30g tubes sufficient for each participants to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- 3% Menthol: 3% menthol gel was supplied in 30g tubes sufficient for each participants to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- Placebo: Placebo with 0.09% methanol gel was supplied in 30g tubes sufficient for each participants to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
Hours | 92.50 [0.2 to 203.8] | 76.83 [0.2 to 184.1] | 72.00 [0.2 to 203.5] | 93.50 [0.2 to 203.0]
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium+3% Menthol vs Placebo; Test type: Superiority or Other; p = 0.6918, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 0.93, 95% CI 2-sided [0.67 to 1.31] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: 1% Diclofenac Sodium+3% Menthol vs 3% Menthol; Test type: Superiority or Other; p = 0.2389, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.23, 95% CI 2-sided [0.87 to 1.73] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 1% Diclofenac Sodium+3% Menthol vs 1% Diclofenac Sodium; Test type: Superiority or Other; p = 0.9817, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.00, 95% CI 2-sided [0.74 to 1.37] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Time of Onset of Cooling Sensation (TOCS)
Description: Time of onset of cooling sensation measured by time when subjects reported to have a 'cooling effect as an enhancement of pain relief'. To assess this endpoint, participants were asked at 10, 30 minutes and at 1, 4, 6 hours post first dose "Do you feel a cooling sensation at the injured ankle from the study gel?
Time Frame: up to 6 hours
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
Hours | 0.17 [0.17 to 6.0] | 0.17 [0.17 to 6.0] | 0.17 [0.17 to 6.0] | 0.17 [0.17 to 6.0]
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium+3% Menthol vs Placebo; Test type: Superiority or Other; p = 0.7003, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.06, 95% CI 2-sided [0.79 to 1.43] — Cox proportional hazard ratio of survival time, i.e. time to cooling sensation. The 95% confidence intervals of cox proportional hazard ratio
Statistical Analysis 2: Comparison: 1% Diclofenac Sodium+3% Menthol vs 3% Menthol; Test type: Superiority or Other; p = 0.9565, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.01, 95% CI 2-sided [0.75 to 1.35] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: 1% Diclofenac Sodium+3% Menthol vs 1% Diclofenac Sodium; Test type: Superiority or Other; p = 0.6216, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.07, 95% CI 2-sided [0.82 to 1.40] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: TOTPAR was calculated as sum of the products of PRS with time interval from one time point to the other. PRS was measured at each time point on a scale: 0= No pain relief, 1= A little or perceptible pain relief, 2= Meaningful pain relief, 3= A lot of relief, 4= Complete relief. The possible range of TOTPAR for 0-6 hours was from 0 to 24, for 0-12 hours was from 0 to 48, for 0-24 hours was from 0 to 96, for 0-72 hours was from 0 to 288, for 24-72 hours was from 0 to 192 and for 0-168 hours was from 0 to 672.
Time Frame: Baseline to 168 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: PRS Score (0 - 4 scale)
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
PRS Score (0 - 4 scale)
  0-6 hours | 2.81 (3.162) | 2.64 (2.902) | 3.27 (3.176) | 2.75 (3.184)
  0-12 hours | 6.86 (6.125) | 6.81 (6.178) | 8.02 (7.045) | 6.35 (6.732)
  0- 24 hours | 16.04 (12.048) | 16.14 (12.479) | 18.85 (14.517) | 15.71 (13.146)
  0-72 hours | 60.14 (37.867) | 61.24 (35.877) | 66.69 (40.360) | 58.75 (41.724)
  24-72 hours | 44.10 (29.344) | 45.11 (26.431) | 47.84 (29.102) | 43.04 (31.570)
  0-168 hours | 172.97 (98.838) | 170.73 (97.187) | 184.17 (102.787) | 174.00 (94.917)

11. Secondary Outcome: Skin Temperature
Description: Skin temperature was measured by thermal imaging.
Time Frame: At 10, 30, 60 minutes, 4 and 6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degree celsius (°C)
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 11 | 10 | 6 | 6
degree celsius (°C)
  At 10 min. | 27.69 (3.706) | 29.31 (2.610) | 29.92 (2.118) | 30.93 (2.842)
  At 30 min. | 28.26 (3.161) | 29.81 (2.595) | 30.50 (2.117) | 31.47 (3.386)
  At 60 min. | 28.64 (2.986) | 30.74 (2.781) | 30.22 (2.388) | 31.78 (3.213)
  At 240 min. | 30.52 (2.880) | 31.26 (2.981) | 31.15 (3.221) | 31.57 (2.700)
  At 360 min. | 31.02 (2.951) | 31.53 (3.299) | 31.27 (3.925) | 32.07 (3.482)

12. Secondary Outcome: Ankle Swelling
Description: Ankle swelling measured by "figure of eight" method of injured ankle.
Time Frame: Day 1 (baseline), 3, and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
Millimeters
  At Day 1 | 573.9 (57.77) | 573.6 (50.20) | 577.1 (55.35) | 576.1 (50.19)
  At Day 3 | 566.2 (57.03) | 566.9 (49.55) | 567.0 (56.48) | 565.4 (52.67)
  At Day 7 | 558.3 (56.02) | 558.8 (46.37) | 558.4 (56.88) | 557.0 (50.85)

13. Secondary Outcome: Time to Complete Recovery
Description: Time to complete recovery measured as the day with complete relief of ankle pain (Participant-rated NRS scores were 0 for pain intensity at rest and pain) and swelling (Participants did not have any apparent swelling nor experience any pain or limitation of movement of the injured ankle as determined by the Principal Investigator or designee during the course of an ankle exam).
Time Frame: up to 240 hours
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 117 | 112 | 77 | 75
Hours | 240.00 [17.0 to 240.0] | 240.00 [48.2 to 240.0] | 240.00 [53.2 to 240.0] | 240.00 [145.5 to 240.0]
Statistical Analysis 1: Comparison: 1% Diclofenac Sodium+3% Menthol vs Placebo; Test type: Superiority or Other; p = 0.0408, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 2.43, 95% CI 2-sided [1.04 to 5.70] — Cox proportional hazard ratio of survival time, i.e. time to complete pain relief. The 95% confidence intervals of cox proportional hazard ratio
Statistical Analysis 2: Comparison: 1% Diclofenac Sodium+3% Menthol vs 3% Menthol; Test type: Superiority or Other; p = 0.4507, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.31, 95% CI 2-sided [0.65 to 2.65] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 1% Diclofenac Sodium+3% Menthol vs 1% Diclofenac Sodium; Test type: Superiority or Other; p = 0.3150, chi-square test of survival analysis — P-value from chi-square test of survival analysis; Cox proportional hazard ratio = 1.38, 95% CI 2-sided [0.73 to 2.61] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Patient's Global Assessment in Response to Treatment (PGART)
Description: PGART was measured at the end of study in a scale from 0-4 (Where: 0- Poor; 1- Fair; 2- Good; 3- Very Good; 4- Excellent)
Time Frame: up to Day 10
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | 1% Diclofenac Sodium+3% Menthol | 1% Diclofenac Sodium | 3% Menthol | Placebo
Number analyzed (Participants) | 115 | 111 | 75 | 75
Participants
  Poor=0 | 3 (0.948) | 13 (1.051) | 6 (1.040) | 9 (1.084)
  Fair=1 | 24 | 20 | 12 | 14
  Good=2 | 44 | 46 | 26 | 27
  Very Good=3 | 35 | 26 | 26 | 21
  Excellent=4 | 9 | 6 | 5 | 4

ADVERSE EVENTS:
Time Frame: Up to 3 weeks of administration of investigational product
Groups:
- 1% Diclofenac Sodium Plus 3% Menthol: 1% diclofenac sodium plus 3% menthol gel supplied in 30 gram (g) tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- 1% Diclofenac Sodium Plus 0.09% Menthol: 1% diclofenac sodium plus 0.09% menthol gel supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
- Placebo With 0.09% Menthol Gel: Placebo with 0.09% menthol gel supplied in 30g tubes sufficient for each participant to apply 4g of gel to the injured ankle region four times daily for up to 10 days.
Arm/Group | 1% Diclofenac Sodium Plus 3% Menthol | 1% Diclofenac Sodium Plus 0.09% Menthol | 3% Menthol | Placebo With 0.09% Menthol Gel
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/112 | 0/77 | 0/75
Other Adverse Events (participants affected / at risk) | 43/117 | 26/112 | 22/77 | 17/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Diclofenac Sodium Plus 3% Menthol (N=117) | 1% Diclofenac Sodium Plus 0.09% Menthol (N=112) | 3% Menthol (N=77) | Placebo With 0.09% Menthol Gel (N=75)
APPLICATION SITE DRYNESS (General disorders) | 15 | 7 | 3 | 4
APPLICATION SITE PAIN (General disorders) | 7 | 0 | 2 | 1
APPLICATION SITE PRURITUS (General disorders) | 5 | 3 | 1 | 1
APPLICATION SITE ERYTHEMA (General disorders) | 4 | 1 | 2 | 0
APPLICATION SITE ECZEMA (General disorders) | 2 | 0 | 0 | 0
APPLICATION SITE DISCOLOURATION (General disorders) | 1 | 0 | 0 | 0
APPLICATION SITE RASH (General disorders) | 1 | 0 | 0 | 0
APPLICATION SITE REACTION (General disorders) | 1 | 0 | 0 | 0
APPLICATION SITE VESICLES (General disorders) | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0 | 0
NECROSIS (General disorders) | 1 | 0 | 0 | 0
APPLICATION SITE BURN (General disorders) | 0 | 0 | 1 | 0
APPLICATION SITE HYPERSENSITIVITY (General disorders) | 0 | 1 | 0 | 0
APPLICATION SITE SWELLING (General disorders) | 0 | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 | 10 | 10 | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 7 | 4 | 3 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 6 | 2 | 3 | 1
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
SKIN WRINKLING (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 4 | 2 | 4 | 3
BURNING SENSATION (Nervous system disorders) | 1 | 0 | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
PYODERMA (Infections and infestations) | 1 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
MUSCLE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
BONE SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.